CLINICAL TRIAL: NCT06935565
Title: Clinical Performance of the Asqelio™ Trifocal Diffractive Intraocular Lens
Status: Completed | Type: Observational
Sponsor: AST Products, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: ASQT012022
Record Dates: First submitted 2025-02-27; First posted 2025-04-20 (Actual); Last update posted 2025-04-20 (Actual); Status verified 2025-04

CONDITIONS: Cataract
Keywords: multifocal IOL; optical quality; visual performance
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Trifocal: Patients implanted bilterally with Asqelio Trifocal IOL
  Interventions: Other: Trifocal IOL implantation

INTERVENTIONS:
Other: Trifocal IOL implantation — Patients were implanted bilaterally with Asqelio Trifocal IOL 270±90 days before study visit

SUMMARY:
The goal of this observational study is to evaluate whether the Asqelio™ Trifocal intraocular lens (IOL) can improve refractive outcomes and optical quality in patients (aged ≥45 years) undergoing cataract surgery or clear lens exchange, including both male and female participants. The main questions it aims to answer are:

* Does the Asqelio™ Trifocal IOL provide accurate refractive correction with minimal residual refractive error?
* Does the lens reduce light distortion and provide good visual acuity at multiple distances (far, intermediate, near)?

Researchers will not use a comparison group, as this is a post-marketing, single-arm observational study.

Participants will undergo bilateral implantation of the Asqelio™ Trifocal IOL during cataract or lens replacement surgery and attend a study follow-up exam approximately 270±90 days post-surgery.

Complete evaluations including:

* Manifest refraction testing
* Uncorrected and corrected visual acuity at far, intermediate, and near distances
* Binocular defocus curve analysis
* Contrast sensitivity testing
* Light distortion analysis using a Light Distortion Analyzer
* Patient-reported outcomes via the Catquest-9SF and visual symptoms questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Patients 50 years of age or older undergoing cataract surgery by phacoemulsification and binocular IOL implant AsqelioTM Trifocal TFLIO130C
* Independence of use of glasses after surgery.
* IOL power between +5.0D and +34.0D
* Transparent intraocular media except for cataracts in both eyes.
* Potential postoperative visual acuity of 20/25 or better.

Exclusion Criteria:

* Preoperative corneal astigmatism greater than 1.0D
* Previous corneal surgery or trauma.
* Irregular cornea (e.g. keratoconus)
* Choroidal hemorrhage
* Microphtalmos
* Severe corneal dystrophy
* Uncontrolled or medically controlled glaucoma
* Clinically significant macular changes
* Concomitant severe eye disease
* Non-age-related cataract
* Severe optic nerve atrophy
* Diabetic retinopathy
* Proliferative diabetic retinopathy
* Amblyopia
* Extremely shallow anterior camera
* Severe chronic uveitis
* Pregnant or nursing
* Rubella
* Mature/dense cataract that makes it difficult to examine the eye fundus preoperatively.
* Previous retinal detachment
* Concurrent participation in other research with drugs or clinical devices

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients of usual clinical practice who have undergone conventional cataract surgery by phacoemulsification and wish to eliminate their refractive error and correct their presbyopia
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2022-09-02 (Actual); Primary Completion 2023-06-15 (Actual); Study Completion 2024-10-14 (Actual)

PRIMARY OUTCOMES:
Residual refraction | 270±90 days after surgery
  Residual refractive error determined by subjective refraction procedures and expressed in diopters of spherical and cylindrical power
Light Distortion Index | 270±90 days from surgery
  The distortion index is calculated as the ratio of the area of points missed by the subject and the total area explored using the Light Distortion Analyzer, and is expressed as a percentage

SECONDARY OUTCOMES:
Visual acuity | 270±90 days after surgery
  The VA with its best correction placed under photopic conditions was determined monocularly at a distance of 4 meters (UDVA and BCDVA), 60 cm (UIVA and BDCIVA), 40 cm (UNVA and BDCNVA), using the optotype of letters Early Treatment Diabetic Retinopathy Study (ETDRS)
Binocular defocus curve | 270±90 days after surgery
  Binocular defocus curve was obtained by varying the stimulus vergence from -4.0 D to +2.0 D in 0.5 D steps with the best correction for distance vision
Contrast sensitivity | 270±90 days after surgery
  The spatial profile of the stimulus was configured to diplay sinusoidal patterns in a circular window with sharp or smoothed edges. The patient's task was to describe the orientation of the stimulus, which changes at random among three options: vertical (grating at 0°), right (15°), or left (-15°), using the Topcon CC-100 instrument
Patient-Reported Outcomes - CATQuest9SF | 270±90 days after surgery
  9-item questionnaire to determine patient activity limitations in daily life due to poor vision used due to its documented responsiveness in cataract surgery. It comprises 9 items with 4 response options, ranging from 4 for "very great difficulty/very dissatisfied" to 1 for "no difficulty/very satisfied", and a "cannot decide" additional option, which is treated as missing data. The questionnaire responses were scored using the Likert scale, from 1 for no difficulty/very satisfied, to 4 for very great difficulty/very dissatisfied.
Patient-Reported Outcomes - Visual symptoms | 270±90 days after surgery
  A visual symptoms questionnaire explores the frequency, intensity and bothersome of 10 different and common visual symptoms. These symptoms are: Glare, Haloes, Starbursts, Foggy vision, Blurred vision, Distortion, Double vision, Fluctuation in vision, Difficulty focusing, and Difficulty judging distances or depth. A simulated image is shown to the patient to aid in the description of each of the symptoms, and they are asked to respond with 4 response options to the frequency of the symptoms, from 1 for "Never" to 4 "Very often", the intensity of the symptom, from 1 for "None" to 4 for "Severe", and the level of bothersome of the symptom, from 1 for "None" to 4 for "A lot". The scoring of these responses ranges from 0 for Never/None to 3 for Very Often/Severe/A lot

CONTACTS AND LOCATIONS:
Locations (1):
- Clinica Baviera, Seville, Seville, Spain

IPD SHARING:
Plan to Share IPD: Undecided